CLINICAL TRIAL: NCT02973789
Title: LUNAR: Pivotal, Randomized, Open-label Study of Tumor Treating Fields (TTFields) Concurrent With Standard of Care Therapies for Treatment of Stage 4 Non-small Cell Lung Cancer (NSCLC) Following Platinum Failure
Brief Title: Effect of Tumor Treating Fields (TTFields) (150 kHz) Concurrent With Standard of Care Therapies for Treatment of Stage 4 Non-small Cell Lung Cancer (NSCLC) Following Platinum Failure (LUNAR)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NovoCure GmbH (Industry)
Responsible Party: Sponsor
Organization: NovoCure Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF-24
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2024-10-21 (Actual); Status verified 2024-09

CONDITIONS: Nonsmall Cell Lung Cancer; NSCLC
Keywords: Non-Small Cell Lung Cancer; NSCLC; Treatment; Minimal Toxicity; TTFields; TTF; Tumor Treating Fields; Novocure; Docetaxel; PD-1 inhibitor; PD-L1 inhibitor; Immune checkpoint inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immune Checkpoint Inhibitors; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- NovoTTF-200T (Experimental): Patients receive TTFields using the NovoTTF-200T device together with immune checkpoint inhibitors or docetaxel
  Interventions: Device: NovoTTF-200T; Drug: Immune checkpoint inhibitors or docetaxel
- Best Standard of Care (Active Comparator): Patients receive best standard of care with immune checkpoint inhibitors or docetaxel
  Interventions: Drug: Immune checkpoint inhibitors or docetaxel

INTERVENTIONS:
Device: NovoTTF-200T — Patients receive continuous TTFields treatment using the NovoTTF-200T device. TTFields treatment will consist of wearing four electrically insulated electrode arrays on the chest. The treatment enables the patient to maintain regular daily routine.
  Other Name: TTFields
  Drug: Immune checkpoint inhibitors or docetaxel Patients receive standard of care with Immune checkpoint inhibitors or docetaxel
  Other Names: TTFields
  Arms: NovoTTF-200T
Drug: Immune checkpoint inhibitors or docetaxel — Patients receive standard of care with Immune checkpoint inhibitors or docetaxel

SUMMARY:
The study is a prospective, randomized controlled phase III trial aimed to test the efficacy and safety of TTFields, using the NovoTTF-200T device, concurrent with standard therapies for stage 4 NSCLC patients, following progression while on or after platinum based treatment. The device is an experimental, portable, battery operated device for chronic administration of alternating electric fields (termed TTFields or TTF) to the region of the malignant tumor, by means of surface, insulated electrode arrays.

DETAILED DESCRIPTION:
PAST PRE-CLINICAL AND CLINICAL EXPERIENCE:

The effect of the electric fields (TTFields, TTF) has demonstrated significant activity in in vitro and in vivo NSCLC pre-clinical models both as a single modality treatment and in combination with chemotherapies and PD-1 inhibitors. TTFields have been demonstrated to act synergistically with taxanes and have been shown to be additive when combined with PD-1 inhibitors. In addition, TTFields have shown to inhibit metastatic spread of malignant melanoma in in vivo experiment.

In a pilot study, 42 patients with advanced NSCLC who had had tumor progression after at least one line of prior chemotherapy, received pemetrexed together with TTFields (150 kHz) applied to the chest and upper abdomen until disease progression (Pless M., et al., Lung Cancer 2011). The combination was well tolerated and the only device-related adverse event was mild to moderate contact dermatitis. Efficacy endpoints were remarkably high compared to historical data for pemetrexed alone.

In addition, a phase III trial of Optune® (200 kHz) as monotherapy compared to active chemotherapy in recurrent glioblastoma patients showed TTFields to be equivalent to active chemotherapy in extending survival, associated with minimal toxicity, good quality of life, and activity within the brain (14% response rate) (Stupp R., et al., EJC 2012). Finally, a phase III trial of Optune® combined with maintenance temozolomide compared to maintenance temozolomide alone has shown that combined therapy led to a significant improvement in both progression free survival and overall survival in patients with newly diagnosed glioblastoma without the addition of high grade toxicity and without decline in quality of life (Stupp R., et al., JAMA 2015).

DESCRIPTION OF THE TRIAL:

All patients included in this trial are patients with squamous or non-squamous, stage 4 NSCLC who had disease progression on or after receiving platinum based chemotherapy. In addition, all patients must meet all eligibility criteria.

Eligible patients will be randomly assigned to one of two groups:

Patients receive docetaxel or immune checkpoint inhibitor in combination with TTFields using the NovoTTF-100L System.

Patients receive docetaxel or immune checkpoint inhibitor without TTFields. Patients will be randomized at a 1:1 ratio. Baseline tests will be performed in patients enrolled in both arms. If assigned to the NovoTTF-100L group, the patients will be treated continuously with the device until disease progression in the thorax and/or liver according to RECIST or irRECIST (Immune-Related Response Evaluation Criteria In Solid Tumors) (depending if the patient is receiving docetaxel or immune checkpoint inhibitor, respectively).

On both arms, patients who have disease progression according to RECIST or irRECIST (depending if the patient is receiving docetaxel or immune checkpoint inhibitor, respectively) will switch to a third line treatment according to local practice.

SCIENTIFIC BACKGROUND:

Electric fields exert forces on electric charges similar to the way a magnet exerts forces on metallic particles within a magnetic field. These forces cause movement and rotation of electrically charged biological building blocks, much like the alignment of metallic particles seen along the lines of force radiating outwards from a magnet.

Electric fields can also cause muscles to twitch and if strong enough may heat tissues. TTFields are alternating electric fields of low intensity. This means that they change their direction repetitively many times a second. Since they change direction very rapidly (150 thousand times a second), they do not cause muscles to twitch, nor do they have any effects on other electrically activated tissues in the body (brain, nerves and heart). Since the intensities of TTFields in the body are very low, they do not cause heating.

The breakthrough finding made by Novocure was that finely tuned alternating fields of very low intensity, now termed TTFields (Tumor Treating Fields), cause a significant slowing in the growth of cancer cells. Due to the unique geometric shape of cancer cells when they are multiplying, TTFields cause electrically-charged cellular components of these cells to change their location within the dividing cell, disrupting their normal function and ultimately leading to cell death. In addition, cancer cells also contain miniature building blocks which act as tiny motors in moving essential parts of the cells from place to place. TTFields interfere with the normal orientation of these tiny motors related to other cellular components since they are electrically-charged as well. As a result of these two effects, tumor cell division is slowed, results in cellular death or reverses after continuous exposure to TTFields.

Other cells in the body (normal healthy tissues) are affected much less than cancer cells since they multiply at a much slower rate if at all. In addition TTFields can be directed to a certain part of the body, leaving sensitive areas out of their reach. Finally, the frequency of TTFields applied to each type of cancer is specific and may not damage normally dividing cells in healthy tissues.

In conclusion, TTFields hold the promise of serving as a brand new treatment for NSCLC with very few side effects.

ELIGIBILITY:
Inclusion Criteria:

1. 22 years of age and older (some regional variations to inclusion age exist)
2. Life expectancy of ≥ 3 months
3. Histological diagnosis of squamous or non-squamous, inoperable, metastatic NSCLC
4. Diagnosis of radiological progression while on or after first platinum-based systemic therapy administered for advanced or metastatic disease.

   1. Patients who received adjuvant or neoadjuvant platinum-based chemotherapy (after surgery and/or radiation therapy) and developed metastatic disease within 6 months of completing therapy are eligible.
   2. Patients with metastatic disease more than 6 months after adjuvant or neoadjuvant platinum-based chemotherapy, who also subsequently progressed during or after a platinum- based regimen given to treat the advanced or metastatic disease, are eligible.
   3. Patients should not receive any systemic therapy after platinum failure before enrollment into the study. Maintenance therapy after platinum based therapy and prior to progression is allowed.
5. ECOG Score of 0-2
6. Assigned by the physician to receive either docetaxel or immune checkpoint inhibitor per standard of care regimen
7. Able to operate the NovoTTF-200T device independently or with the help of a caregiver
8. Signed informed consent for the study protocol

Exclusion Criteria:

1. Metastases to central nervous system (CNS) with clinical symptoms or evidence of new metastases to CNS during screening. Patients who previously received treatments for the metastases to CNS, are stable and meet the following requirements are allowed to be enrolled:

   1. The patients are neurologically returned to baseline (except for residual signs or symptoms related to CNS treatment).
   2. No treatment for the metastases to CNS during the screening period (e.g. surgery, radiotherapy, corticosteroid therapy- prednisone > 10 mg/day or equivalent).
   3. No progress in CNS lesions as indicated by MRI within 14 days prior to randomization.
   4. No meningeal metastasis or spinal cord compression.
2. Patients planned to receive immune checkpoint inhibitor with contra-indications to receive immunotherapy
3. Patients planned to receive docetaxel with contra-indications to receive docetaxel
4. Severe comorbidities:

   1. Clinically significant (as determined by the investigator) hematological, hepatic and renal dysfunction, defined as: Neutrophil count < 1.5 x 10^9/L and platelet count < 100 x 10^9/L; bilirubin > 1.5 x ULN; AST and/or ALT > 2.5 x ULN or > 5 x ULN if patient has documented liver metastases; and serum creatinine > 1.5 x ULN
   2. History of significant cardiovascular disease unless the disease is well controlled. Significant cardiac disease includes second/third degree heart block; significant ischemic heart disease; poorly controlled hypertension; congestive heart failure of the New York Heart Association (NYHA) Class II or worse (slight limitation of physical activity; comfortable at rest, but ordinary activity results in fatigue, palpitation or dyspnea)
   3. History of arrhythmia that is symptomatic or requires treatment. Patients with atrial fibrillation or flutter controlled by medication are not excluded from participation in the trial
   4. History of pericarditis
   5. History of interstitial lung disease
   6. History of cerebrovascular accident (CVA) within 6 months prior to randomization or that is not stable
   7. Active infection or serious underlying medical condition that would impair the ability of the patient to received protocol therapy
   8. History of any psychiatric condition that might impair patient's ability to understand or comply with the requirements of the study or to provide consent
   9. Any other malignancy requiring anti-tumor treatment in the past three years, excluding treated stage I prostate cancer, in situ cervical cancer, in situ breast cancer and non-melanomatous skin cancer
5. Concurrent treatment with other experimental treatments for NSCLC while on the study
6. Implantable electronic medical devices (e.g. pacemaker, defibrillator) in the upper torso
7. Known allergies to medical adhesives or hydrogel
8. Pregnancy or breast-feeding (patients with reproductive potential must use effective contraception methods throughout the entire study period, as determined by their investigator/gynecologist)
9. Admitted to an institution by administrative or court order

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2016-12; Primary Completion 2024-09-24 (Actual); Study Completion 2024-10-09 (Actual)

PRIMARY OUTCOMES:
Overall survival of patients treated with TTFields + docetaxel or immune checkpoint inhibitors vs. docetaxel or immune checkpoint inhibitors alone (superiority analysis) | 4 years

SECONDARY OUTCOMES:
Overall survival of patients treated with TTFields + docetaxel vs. docetaxel alone (superiority analysis) | 4 years
Overall survival of patients treated with TTFields + immune checkpoint inhibitors vs. immune checkpoint inhibitors alone (superiority) | 4 years
Overall Survival of patients treated with TTFields + docetaxel Vs. immune checkpoint inhibitors alone (non-inferiority analysis) | 4 years
Progression-free survival of patients treated with docetaxel or immune checkpoint inhibitors + TTFields vs. docetaxel or immune checkpoint inhibitors alone, based on RECIST Criteria | 4 years
Overall radiological response rate (based on RECIST criteria) of patients treated with docetaxel or Immune checkpoint inhibitors + TTFields vs. docetaxel or immune checkpoint inhibitors alone. | 4 years
Quality of life using the EORTC QLQ C30 questionnaire with LC13 addendum | 4 years
Analyses of the effects of NovoTTF-200T with each type of immune checkpoint inhibitor on overall survival and progression free survival | 4 years
Analysis of the effects of NovoTTF-200T on overall survival and progression free survival within each histological subgroup (squamous and non-squamous) | 4 years
The effect of treatment compliance with NovoTTF-200T on overall survival and progression free survival outcomes | 4 years
Adverse events, severity and frequency based on Common Terminology Criteria for Adverse Events (CTCAE) V4.03 | 4 years

CONTACTS AND LOCATIONS:
Locations (124):
- United States (73):
  - Central Alabama Research, Birmingham, Alabama
  - Ironwood Cancer & Research Center, Chandler, Arizona
  - Cancer Center at St. Joseph Hospital and Medical Center, Phoenix, Arizona
  - Beverly Hills Cancer Center, Beverly Hills, California
  - California Cancer Associates for Research and Excellence, Inc. cCARE, Fresno, California
  - St. Joseph Heritage Healthcare, Fullerton, California
  - Saddleback Memorial Medical Center, Laguna Hills, California
  - Redlands Community Hospital (Emad Ibrahim, MD, Inc.), Redlands, California
  - Dignity Health - Mercy Cancer Centers, Sacramento, California
  - Sutter Institute for Medical Research, Sacramento, California
  - Innovative Clinical Research Institute, Whittier, California
  - Banner MD Anderson Cancer Center at North Colorado Medical Center, Greeley, Colorado
  - Associated Neurologists of Southern CT, P.C., Fairfield, Connecticut
  - Washington Cancer Institute at MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - GenesisCare USA, Jacksonville, Florida
  - Miami Cancer Institute, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Adult Oncology Research, Orlando, Florida
  - BRCR Medical Center INC, Plantation, Florida
  - University of Illinois Cancer Center, Chicago, Illinois
  - Illinois CancerCare, P.C., Peoria, Illinois
  - Southern Illinois University, School of Medicine, Simmons Cancer Institute at SIU, Springfield, Illinois
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - University of Kansas Cancer Center, Westwood, Kansas
  - Norton Cancer Institute, Louisville, Kentucky
  - University Medical Center, Inc; DBA University of Louisville, Louisville, Kentucky
  - LSU Health Sciences Center -New Orleans, New Orleans, Louisiana
  - Tulane Cancer Center, New Orleans, Louisiana
  - CHRISTUS Health, Shreveport, Louisiana
  - Central Maine Medical Center, Lewiston, Maine
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Tufts Medical Center, Division of Hematology and Oncology, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Clinical Oncology Associates, Farmington Hills, Michigan
  - Detroit Clinical Research Center, Farmington Hills, Michigan
  - Saint Joseph Mercy Health System, Ypsilanti, Michigan
  - HealthPartners Institute, Regions Cancer Care Center, Saint Paul, Minnesota
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - CHI Health Research Center, Omaha, Nebraska
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - OptumCare Cancer Care, Las Vegas, Nevada
  - Renown Regional Medical Center Institute for Cancer, Reno, Nevada
  - Presbyterian Cancer Center, Albuquerque, New Mexico
  - New York-Presbyterian/Queens Radiation Oncology, Flushing, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Stony Brook Cancer Center, Stony Brook, New York
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - W.G. Bill Hefner VA Med Center, Salisbury, North Carolina
  - Piedmont Radiation Oncology, PA, Winston-Salem, North Carolina
  - Summa Health, Akron, Ohio
  - Toledo Clinic Cancer Center, Toledo, Ohio
  - Vita Medical Associates, P.C., Bethlehem, Pennsylvania
  - Geisinger Cancer Institute, Danville, Pennsylvania
  - UT/Erlanger Oncology & Hematology, Chattanooga, Tennessee
  - Texas Oncology - Amarillo, Amarillo, Texas
  - Texas Oncology - Arlington, Arlington, Texas
  - Christus Health Spohn Ministry, Corpus Christi, Texas
  - Dallas VA Medical Center, Dallas, Texas
  - Texas Oncology- Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Oncology Consultants, P.A., Houston, Texas
  - Texas Oncology-McKinney, McKinney, Texas
  - Texas Oncology - Paris, Paris, Texas
  - Texas Oncology- Plano West, Plano, Texas
  - Baylor Scott & White Health/McClinton Cancer Center, Waco, Texas
  - Texas Oncology-Waco, Waco, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Overlake Medical Center & Clinics, Bellevue, Washington
  - UW Carbone Cancer Center, Madison, Wisconsin
- Medical University Salzburg, State Hospital, University hospital for internal medicine III / PMU, Salzburg, Austria
- Belgium (3):
  - Institut Jules Bordet - Department of Intensive Care and Thoracic Oncology, Brussels
  - Clinique André Renard Herstal Oncologie, Herstal
  - AZ Sint Maarten, Mechelen
- Complex Oncology Center (COC) - Plovdiv EOOD,, Plovdiv, Bulgaria
- Canada (3):
  - McGill University Health Centre, Montreal, Quebec
  - Centre intégré universitaire de santé et de services sociaux de l'Estrie - Centre Hospitalier Universitaire de Sherbrooke (CIUSSS de l'Estrie - CHUS), Sherbrooke, Quebec
  - Allan Blair Cancer Center, Regina, Saskatchewan
- China (8):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Affiliated Cancer Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - PKUCare Luzhong Hospital, Zibo, Shandong
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Sun Yat-sen University Cancer Center, Guangzhou
- University Hospital Centre Zagreb, Zagreb, Croatia
- Czechia (3):
  - General University Hospital in Prague, Prague
  - Thomayerova Nemocnice Dept. of Pneumology, Prague
  - Vitkovicka nemocnice, Vítkovice
- France (6):
  - Centre Hospitalier de Beauvais, Beauvais
  - INSTITUT BERGONIE Centre Régional de Lutte Contre le Cancer, Bordeaux
  - Groupe Hospitalier Bretagne Sud, Lorient
  - CHU Caremeau Service de Pneumologie, Nîmes
  - AH-HP Hôpital Saint Louis, Paris
  - Centre Hospitalier de Saint-Quentin Service de pneumologie, Saint-Quentin
- Universitätsklinikum Halle - Universitätsklinik und Poliklinik für Innere Medizin IV, Halle, Germany
- Queen Mary Hospital, Hong Kong, Hong Kong
- Tolna County, Balassa Janos Hospital, Department of oncology, Szekszárd, Hungary
- Italy (4):
  - ASL 3, Ospedale Villa Scassi, Genova
  - IRCCS - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Meldola
  - UOC Oncologia Medica Presidio Ospedaliero di Ravenna AUSL della Romagna, Ravenna
  - Saronno Hospital, Saronno
- Netherlands (2):
  - St Jansdal Ziekenhuis, Harderwijk
  - Erasmus Mc, Rotterdam
- Poland (5):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Centrum Terapii Współczesnej, Lodz
  - MS Clinsearch Specjalistyczny NZOZ, Lublin
  - Clinical Hospital of Przemienienia Pańskiego UM in Poznaniu, Poznan
  - Samodzielny Publiczny Wojewódzki Szpital Zespolony w Szczecinie, Szczecin
- Serbia (2):
  - Bezanijska kosa Clinical Hospital Center, Belgrade
  - University Clinical Center Kragujevac, Kragujevac
- Spain (8):
  - Hospital Universitario Arnau de Vilanova, Lleida, Catalonia
  - Hospital Quirón Teknon, Instituto Oncológico Dr. Rosell, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Regional Universitario Carlos Haya Medical Oncology Department, Málaga
  - Hospital Virgen de la Salud, Toledo
  - Hospital Universitari i Politécnic La Fe, Valencia
- Kantonsspital Winterthur Tumorzentrum Winterthur, Winterthur, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kirson ED, Gurvich Z, Schneiderman R, Dekel E, Itzhaki A, Wasserman Y, Schatzberger R, Palti Y. Disruption of cancer cell replication by alternating electric fields. Cancer Res. 2004 May 1;64(9):3288-95. doi: 10.1158/0008-5472.can-04-0083. PMID 15126372
- [Background] Kirson ED, Dbaly V, Tovarys F, Vymazal J, Soustiel JF, Itzhaki A, Mordechovich D, Steinberg-Shapira S, Gurvich Z, Schneiderman R, Wasserman Y, Salzberg M, Ryffel B, Goldsher D, Dekel E, Palti Y. Alternating electric fields arrest cell proliferation in animal tumor models and human brain tumors. Proc Natl Acad Sci U S A. 2007 Jun 12;104(24):10152-7. doi: 10.1073/pnas.0702916104. Epub 2007 Jun 5. PMID 17551011
- [Background] Stupp R, Wong ET, Kanner AA, Steinberg D, Engelhard H, Heidecke V, Kirson ED, Taillibert S, Liebermann F, Dbaly V, Ram Z, Villano JL, Rainov N, Weinberg U, Schiff D, Kunschner L, Raizer J, Honnorat J, Sloan A, Malkin M, Landolfi JC, Payer F, Mehdorn M, Weil RJ, Pannullo SC, Westphal M, Smrcka M, Chin L, Kostron H, Hofer S, Bruce J, Cosgrove R, Paleologous N, Palti Y, Gutin PH. NovoTTF-100A versus physician's choice chemotherapy in recurrent glioblastoma: a randomised phase III trial of a novel treatment modality. Eur J Cancer. 2012 Sep;48(14):2192-202. doi: 10.1016/j.ejca.2012.04.011. Epub 2012 May 18. PMID 22608262
- [Background] Pless M, Droege C, von Moos R, Salzberg M, Betticher D. A phase I/II trial of Tumor Treating Fields (TTFields) therapy in combination with pemetrexed for advanced non-small cell lung cancer. Lung Cancer. 2013 Sep;81(3):445-450. doi: 10.1016/j.lungcan.2013.06.025. Epub 2013 Jul 23. PMID 23891283
- [Background] Kirson ED, Giladi M, Gurvich Z, Itzhaki A, Mordechovich D, Schneiderman RS, Wasserman Y, Ryffel B, Goldsher D, Palti Y. Alternating electric fields (TTFields) inhibit metastatic spread of solid tumors to the lungs. Clin Exp Metastasis. 2009;26(7):633-40. doi: 10.1007/s10585-009-9262-y. Epub 2009 Apr 23. PMID 19387848
- [Background] Giladi M, Schneiderman RS, Voloshin T, Porat Y, Munster M, Blat R, Sherbo S, Bomzon Z, Urman N, Itzhaki A, Cahal S, Shteingauz A, Chaudhry A, Kirson ED, Weinberg U, Palti Y. Mitotic Spindle Disruption by Alternating Electric Fields Leads to Improper Chromosome Segregation and Mitotic Catastrophe in Cancer Cells. Sci Rep. 2015 Dec 11;5:18046. doi: 10.1038/srep18046. PMID 26658786
- [Background] Giladi M, Weinberg U, Schneiderman RS, Porat Y, Munster M, Voloshin T, Blatt R, Cahal S, Itzhaki A, Onn A, Kirson ED, Palti Y. Alternating electric fields (tumor-treating fields therapy) can improve chemotherapy treatment efficacy in non-small cell lung cancer both in vitro and in vivo. Semin Oncol. 2014 Oct;41 Suppl 6:S35-41. doi: 10.1053/j.seminoncol.2014.09.006. Epub 2014 Sep 8. PMID 25213867
- [Background] Stupp R, Taillibert S, Kanner AA, Kesari S, Steinberg DM, Toms SA, Taylor LP, Lieberman F, Silvani A, Fink KL, Barnett GH, Zhu JJ, Henson JW, Engelhard HH, Chen TC, Tran DD, Sroubek J, Tran ND, Hottinger AF, Landolfi J, Desai R, Caroli M, Kew Y, Honnorat J, Idbaih A, Kirson ED, Weinberg U, Palti Y, Hegi ME, Ram Z. Maintenance Therapy With Tumor-Treating Fields Plus Temozolomide vs Temozolomide Alone for Glioblastoma: A Randomized Clinical Trial. JAMA. 2015 Dec 15;314(23):2535-43. doi: 10.1001/jama.2015.16669. PMID 26670971
- [Background] Voloshin T, Kaynan N, Davidi S, Porat Y, Shteingauz A, Schneiderman RS, Zeevi E, Munster M, Blat R, Tempel Brami C, Cahal S, Itzhaki A, Giladi M, Kirson ED, Weinberg U, Kinzel A, Palti Y. Tumor-treating fields (TTFields) induce immunogenic cell death resulting in enhanced antitumor efficacy when combined with anti-PD-1 therapy. Cancer Immunol Immunother. 2020 Jul;69(7):1191-1204. doi: 10.1007/s00262-020-02534-7. Epub 2020 Mar 6. PMID 32144446
- [Derived] Leal T, Kotecha R, Ramlau R, Zhang L, Milanowski J, Cobo M, Roubec J, Petruzelka L, Havel L, Kalmadi S, Ward J, Andric Z, Berghmans T, Gerber DE, Kloecker G, Panikkar R, Aerts J, Delmonte A, Pless M, Greil R, Rolfo C, Akerley W, Eaton M, Iqbal M, Langer C; LUNAR Study Investigators. Tumor Treating Fields therapy with standard systemic therapy versus standard systemic therapy alone in metastatic non-small-cell lung cancer following progression on or after platinum-based therapy (LUNAR): a randomised, open-label, pivotal phase 3 study. Lancet Oncol. 2023 Sep;24(9):1002-1017. doi: 10.1016/S1470-2045(23)00344-3. PMID 37657460